CLINICAL TRIAL: NCT03489850
Title: Withdrawal-Related Dysphoria as a Moderator of Ibudilast for Alcohol Use Disorder
Brief Title: Ibudilast and Withdrawal-Related Dysphoria
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Lara Ray, PhD, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB#17-001741
Record Dates: First submitted 2018-03-08; First posted 2018-04-06 (Actual); Results first posted 2021-10-07 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-10

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — ibudilast

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ibudilast (Active Comparator): 20mg BID Days 1-2 50mg BID Days 3-14
  Interventions: Drug: Ibudilast
- Placebo (Placebo Comparator): Matched to active
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ibudilast — Ibudilast (IBUD) is a neuroimmune modulator that inhibits phosphodiesterase-4 and -10 and macrophage migration inhibitory factor.
  Arms: Ibudilast
Other: Placebo — Placebo is matched to ibudilast active medication.
  Arms: Placebo

SUMMARY:
Alcohol use disorder (AUD) is a prevalent and disabling psychiatric disorder with few, and only moderately efficacious, treatment options. Consequently, the identification of novel treatment targets and the development of rigorous laboratory paradigms to screen and optimize novel therapeutics represents a research priority. Ibudilast (IBUD) is a neuroimmune modulator that inhibits phosphodiesterase-4 and -10 and macrophage migration inhibitory factor. Recently in an AUD sample, IBUD was shown to decrease reactivity to a psychological stressor. Furthermore, IBUD was effective in blunting alcohol reward among participants with greater depressive symptoms, a hallmark symptom of protracted withdrawal. Recently, preclinical research in opiates has demonstrated that drug withdrawal is necessary for microglia activation and neuroinflammation in reward networks, suggesting that IBUD may be most effective among patients who experience withdrawal-related dysphoria. Therefore, this proposed study aims to examine withdrawal-related dysphoria as a moderator of IBUD efficacy in the natural environment measured using Daily Diary Assessment (DDA) approaches. To accomplish this aim, participants meeting criteria for AUD and balanced on the presence of withdrawal-related dysphoria will be enrolled in a double-blinded IBUD trial including consisting of two weeks randomized to medication and DDA assessment. The proposed research aims are:

Aim 1: Test whether IBUD reduces basal negative affect in abstinence, and blunts alcohol-related negative reinforcement. It is hypothesized that IBUD will reduce basal levels of negative affect during alcohol abstinence, and in so doing will interfere with alcohol-induced blunting of negative affectivity as captured during naturalistic drinking episodes.

Aim 2: Test whether IBUD attenuates neural alcohol cue-reactivity. It is hypothesized that IBUD will reduce BOLD activation to alcohol cues in mesocorticolimbic reward circuitry.

Aim 3: Test whether withdrawal-related dysphoria moderates the effects of IBUD. It is hypothesized that IBUD will alleviate basal negative affect, interfere with alcohol-induced negative reinforcement and attenuate BOLD activation to alcohol cues only among participants who experience dysphoria in withdrawal.

Aim 4: Test whether neural activation to alcohol cues is predictive of drinking outcomes. It is hypothesized that individuals with higher mesocorticolimbic activation to alcohol cues will report more drinking in the week following the neuroimaging session.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 21 and 45
2. Meet DSM-5 criteria for current Moderate-to-Severe AUD
3. Current Heavy Drinking (> 14 drinks per week for men; > 7 drinks per week for women), as indicated by self-reported drinking for the 30 days prior to screening
4. Have reliable internet access

Exclusion Criteria:

1. Currently receiving or seeking treatment for AUD*
2. Past year DSM-5 diagnosis of any substance use disorder other than alcohol or nicotine
3. A lifetime diagnosis of schizophrenia, bipolar disorder, or any psychotic disorder
4. Current use of drugs, other than marijuana, verified by a urine toxicology screen*
5. Pregnant, nursing, or refusal to use reliable birth control (if female)*
6. A medical condition that may interfere with safe participation (e.g., unstable cardiac, renal, or liver disease, uncontrolled hypertension, diabetes, or AST, ALT, or GGT ≥ 3 times upper normal limit)
7. Self-reported recent (i.e. past 30 day) use of medications that are contraindicated with ibudilast*
8. Non-removable ferromagnetic objects in body
9. Claustrophobia
10. Serious head injury or prolonged period of unconsciousness (>30 minutes)

    * Participants who meet these criteria at any point during the course of the study (i.e. after randomization) will be withdrawn from the study for safety purposes.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lara A Ray, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ray LA, Bujarski S, Shoptaw S, Roche DJ, Heinzerling K, Miotto K. Development of the Neuroimmune Modulator Ibudilast for the Treatment of Alcoholism: A Randomized, Placebo-Controlled, Human Laboratory Trial. Neuropsychopharmacology. 2017 Aug;42(9):1776-1788. doi: 10.1038/npp.2017.10. Epub 2017 Jan 16. PMID 28091532
- [Derived] Burnette EM, Ray LA, Irwin MR, Grodin EN. Ibudilast attenuates alcohol cue-elicited frontostriatal functional connectivity in alcohol use disorder. Alcohol Clin Exp Res. 2021 Oct;45(10):2017-2028. doi: 10.1111/acer.14696. Epub 2021 Sep 29. PMID 34585396

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at an outpatient research clinic in a medical center. Participants were recruited through social media and mass transit advertisements. Initial screening was conducted through telephone interview, with eligible participants invited for an in-person assessment.
Period: Overall Study
Arm/Group | Ibudilast | Placebo
Started | 24 | 28
Completed | 23 | 27
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ibudilast | Placebo | Total
Number analyzed (Participants) | 24 | 28 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.46 (9.24) | 31.07 (7.81) | 32.63 (8.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 18
  Male | 16 | 18 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 7 | 12
  Not Hispanic or Latino | 19 | 21 | 40
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 5 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 5 | 2 | 7
  White | 17 | 12 | 29
  More than one race | 1 | 5 | 6
  Unknown or Not Reported | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 24 | 28 | 52
Education [Mean (Standard Deviation); unit: years] | 15.25 (2.64) | 15.21 (1.75) | 15.23 (2.18)
Withdrawal Related Dysphoria [Count of Participants; unit: Participants] | 9 | 11 | 20
Alcohol Use Disorder Symptom Count [Mean (Standard Deviation); unit: symptoms] | 5.29 (2.37) | 4.86 (2.27) | 5.06 (2.30)
Alcohol Use Disorder Identification Test Total Score [Mean (Standard Deviation); unit: score on scale] — The AUDIT has 10 questions and the possible responses to each question are scored 0, 1, 2, 3 or 4, with the exception of questions 9 and 10 which have possible responses of 0, 2 and 4. The range of possible scores is from 0 to 40 where 0 indicates an abstainer who has never had any problems from alcohol. A score of 1 to 7 suggests low-risk consumption according to World Health Organization (WHO) guidelines. Scores from 8 to 14 suggest hazardous or harmful alcohol consumption and a score of 15 or more indicates the likelihood of alcohol dependence (moderate-severe alcohol use disorder).
  score on scale | 16.38 (5.90) | 16.71 (6.42) | 16.56 (6.12)
Alcohol Dependence Scale Total Score [Mean (Standard Deviation); unit: score on scale] — Total scores can range from 0-47. A score of 0 indicates no symptoms. Scores from 1-13 indicate low level of dependence. Scores from 14-21 indicate intermediate levels of dependence. Scores from 22-30 indicate a substantial level of dependence. Scores above 30 indicate a severe level of dependence.
  score on scale | 13.00 (6.10) | 12.07 (7.01) | 12.50 (6.56)
Penn Alcohol Craving Scale Total Score [Mean (Standard Deviation); unit: score] — The PACS is a five-item, self-report measure that includes questions about the frequency, intensity, and duration of craving, the ability to resist drinking, and asks for an overall rating of craving for alcohol for the previous week. Scores can range from 0-30. A score of 0 indicates no craving for alcohol. Higher scores indicate higher craving for alcohol.
  score | 12.79 (5.14) | 12.11 (7.04) | 12.43 (6.18)
Obsessive Compulsive Drinking Scale Total Score [Mean (Standard Deviation); unit: score] — The Obsessive Compulsive Drinking Scale (OCDS) is a 14-item self-rating instrument that provides a total score that measures some cognitive aspects of alcohol craving. The total score range is from 0-40, with higher scores indicating greater severity of AUD. An OCDS total score of 7 and above discriminates between social drinkers and alcohol dependent drinkers, with a sensitivity of 93% and a specificity of 98%.
  score | 14.54 (6.05) | 13.93 (8.07) | 14.21 (7.15)
Reasons for Heavy Drinking Questionnaire - Reinforcing [Mean (Standard Deviation); unit: score] — The Reasons for Heavy Drinking Questionnaire is a brief assessment of motivations for heavy alcohol use. The Reinforcing sub-scale measures the tendency to drink for hedonic (positive reinforcement) and stress relief (negative reinforcement) motivations. Items 1-3 make up the reinforcement sub-scale. Scores range from 0-30. Higher scores indicate more endorsement of drinking motivation for reinforcement.
  score | 23.29 (3.51) | 22.82 (4.88) | 23.04 (4.27)
Reasons for Heavy Drinking Questionnaire - Normalizing [Mean (Standard Deviation); unit: score] — The Reasons for Heavy Drinking Questionnaire is a brief assessment of motivations for heavy alcohol use. The Normalizing sub-scale measures the tendency to drink to feel normal ore avoid withdrawal symptoms. Items 4-6 make up the reinforcement sub-scale. Scores range from 0-30. Higher scores indicate more endorsement of drinking motivation to feel normal.
  score | 9.67 (7.10) | 8.29 (7.34) | 8.92 (7.20)
Total Drinks [Mean (Standard Deviation); unit: drinks over prior 30 days] — Total drinks measures the number of total standard alcoholic drinks consumed as reported on the 30-day Timeline Followback Interview (TLFB).
  drinks over prior 30 days | 122.89 (64.58) | 114.9 (108.72) | 118.20 (90.32)
Drinking Days [Mean (Standard Deviation); unit: number of days in the prior 30 days] — Drinking days measures the number of days an alcohol drink was consumed as reported on the 30-day Timeline Followback Interview (TLFB).
  number of days in the prior 30 days | 22.21 (6.87) | 20.25 (6.51) | 21.15 (6.68)
Drinks Per Day [Mean (Standard Deviation); unit: average drinks over prior 30 days] — Drinks per day measures the number of total standard alcoholic drinks consumed divided by 30 days (average number of drinks per day over 30 days) as reported on the 30-day Timeline Followback Interview (TLFB).
  average drinks over prior 30 days | 4.10 (2.15) | 3.81 (3.62) | 3.94 (3.01)
Drinks Per Drinking Day [Mean (Standard Deviation); unit: drinks] | 5.70 (2.58) | 5.34 (3.57) | 5.51 (3.13)
Heavy Drinking Days [Mean (Standard Deviation); unit: number of heavy drinking days] — Heavy drinking days measures the number of days an individual met heavy drinking standards as reported on the 30-day Timeline Followback Interview (TLFB). Heavy drinking is defined by the National Institute on Alcohol Abuse and Alcoholism (NIAAA) as ≥5 drinks/day for men and ≥4 drinks/day for women.
  number of heavy drinking days | 10.79 (8.29) | 8.68 (8.04) | 9.65 (8.15)
Cigarette Smokers [Count of Participants; unit: Participants] | 11 | 14 | 25
Fagerstrom Test for Nicotine Dependence Score [Mean (Standard Deviation); unit: score on scale] — The Fagerstrom Test for Nicotine Dependence is summed to yield a total score of 0-10. The higher the total Fagerström score, the more intense is the patient's physical dependence on nicotine.
  score on scale | 2.82 (2.82) | 1.07 (1.54) | 1.96 (2.27)
Total Cigarettes [Mean (Standard Deviation); unit: number of cigarettes smoked prior 30 day] — Total cigarettes measures the number of total cigarettes smoked as reported on the 30-day Timeline Followback Interview (TLFB).
  number of cigarettes smoked prior 30 day | 52.28 (79.85) | 133.07 (205.78) | 102.44 (197.18)
Cigarettes Per Day [Mean (Standard Deviation); unit: cigarettes] | 7.39 (8.70) | 5.06 (6.76) | 6.14 (7.73)
THC+ Urine [Count of Participants; unit: Participants] | 7 | 8 | 15
Cannabis Days [Mean (Standard Deviation); unit: number of days used in prior 30 days] — Cannabis days measures the number of days cannabis was used as reported on the 30-day Timeline Followback Interview (TLFB). Cannabis use was assessed by a binary yes or no for each day.
  number of days used in prior 30 days | 11.38 (9.99) | 8.15 (8.24) | 9.64 (9.14)
Beck Depression Inventory-II Total Score [Mean (Standard Deviation); unit: score] — The Beck Depression Inventory-II is a 21-item self-administered survey which is scored on a scale of 0-3 in a list of four statements arranged in increasing severity about a particular symptom of depression. The scores are summed to give a total score. Scores of 0-13 indicate minimal symptoms of depression; scores of 14-19 indicate mild symptoms of depression; scores of 20-28 indicate moderate symptoms of depression; and scores of 29-63 indicate severe symptoms of depression;
  score | 12.42 (8.47) | 8.64 (7.2) | 10.38 (8.27)

OUTCOME MEASURES:

1. Primary Outcome: Negative Affect
Description: Negative affect as measured by self-reported ratings of "Downhearted", "Discouraged", "Uneasy", and "Anxious". Each item was rated on a scale from 0 (not at all) to 4 (extremely). The 4 items were summed for the total negative affect score for each day, ranging from 0 - 16. Higher scores indicate more negative mood.
Time Frame: Assessed through daily prompts throughout the 2-week study period.
Measure: Least Squares Mean (Standard Error); unit: units
Arm/Group | Ibudilast | Placebo
Number analyzed (Participants) | 24 | 28
units | 2.91 (0.55) | 2.47 (0.41)
Statistical Analysis 1: Comparison: Ibudilast vs Placebo; Test type: Superiority; p = .62, Generalized Estimating Equation; Parameter Estimate = 0.34, 95% CI 2-sided [-1.01 to 1.69], Standard Error of Mean 0.69

2. Secondary Outcome: Heavy Drinking
Description: Medication effects on number of heavy drinking days. Heavy drinking is defined by the National Institute on Alcohol Abuse and Alcoholism (NIAAA) as ≥5 drinks/day for men and ≥4 drinks/day for women. Values indicate estimated probability of a heavy drinking day across time for each group.
Time Frame: 14 days
Measure: Number (95% Confidence Interval); unit: predicted probability in percent
Arm/Group | Ibudilast | Placebo
Number analyzed (Participants) | 24 | 28
predicted probability in percent | 24.16 [17.12 to 32.94] | 36.80 [28.43 to 46.05]
Statistical Analysis 1: Comparison: Ibudilast vs Placebo; Test type: Superiority; p < 0.05, Generalized Estimating Equation; Odds Ratio (OR) = 0.55, 95% CI 2-sided [.30 to .98]

3. Secondary Outcome: Any Drinking
Description: Medication effects on number of days where any drinking was reported. . Values indicate estimated probability of a drinking day across time for each group.
Time Frame: 14 days
Measure: Number (95% Confidence Interval); unit: predicted probability in percent
Arm/Group | Ibudilast | Placebo
Number analyzed (Participants) | 24 | 28
predicted probability in percent | 59.25 [47.62 to 69.92] | 63.63 [54.65 to 71.75]
Statistical Analysis 1: Comparison: Ibudilast vs Placebo; Test type: Superiority; p < 0.05, Generalized Estimating Equation; Odds Ratio (OR) = 0.83, 95% CI 2-sided [0.47 to 1.48]

4. Secondary Outcome: Ventral Striatum Activation
Description: Medication effect on alcohol cue-induced ventral striatal activation. Participants completed an fMRI alcohol cue-reactivity paradigm where they viewed pictures of alcoholic beverages, non-alcoholic beverages, blurred images, and a plus sign. The mean percent signal change between the ALC and BEV blocks was extracted from an a priori defined region of interest: bilateral ventral striatum (VS), 6 mm-radius sphere centered at ±12 6 9 in MNI space.
Time Frame: Day 8
Population: Participants were excluded from neuroimaging analyses for the following reasons: participant missed mid-point study visit (n=1, placebo); participant could not be scanned due to COVID-19 safety restrictions (n=1, placebo); participant began scan but ended early due to claustrophobia (n=1, ibudilast); scanner issues prevented the collection of alcohol cue reactivity data (n=1, ibudilast); and participant was found to be not safe for MRI scanning on the day-of the study visit (n=1, ibudilast).
Measure: Mean (Standard Deviation); unit: percent signal change
Arm/Group | Ibudilast | Placebo
Number analyzed (Participants) | 20 | 25
percent signal change | -0.08 (0.20) | 0.14 (0.32)
Statistical Analysis 1: Comparison: Ibudilast vs Placebo; Test type: Superiority; p < 0.05, ANCOVA; F = 7.36

ADVERSE EVENTS:
Time Frame: 2 weeks
Description: Side effects were elicited in open ended fashion and were reviewed by the study physicians (K.M and A.G.). Adverse events were coded using the MedDRA v22.0 coding dictionary. Treatment-emergent adverse events were defined as adverse events that started after the first dose of the study drug or worsened in intensity after the first dose of study drug.
Arm/Group | Ibudilast | Placebo
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/28
Other Adverse Events (participants affected / at risk) | 14/24 | 18/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ibudilast (N=24) | Placebo (N=28)
Nausea (Gastrointestinal disorders) | 6 (6) | 3 (3)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Frequent Bowel Movements (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gut pain (General disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Disorientation (Nervous system disorders) | 1 (1) | 0 (0)
Blurred Vision (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Insomnia (Nervous system disorders) | 2 (2) | 1 (1)
Libido Increased (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 3 (3)
Anxiety (Psychiatric disorders) | 2 (2) | 1 (1)
Grief Reaction (Psychiatric disorders) | 0 (0) | 1 (1)
Irritability (Psychiatric disorders) | 1 (1) | 1 (1)
Cold (Influenza) (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Asthmatic Crisis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cold Sweat (General disorders) | 1 (1) | 0 (0)
Lethargy (General disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-05-10): https://cdn.clinicaltrials.gov/large-docs/50/NCT03489850/Prot_002.pdf
  • Statistical Analysis Plan (2018-05-10): https://cdn.clinicaltrials.gov/large-docs/50/NCT03489850/SAP_003.pdf